CLINICAL TRIAL: NCT01982617
Title: A Randomized, Controlled Trial of Motivational Interviewing Compared to Psychoeducation for Smoking Precontemplators With Severe Mental Illness
Brief Title: Motivational Interviewing Compared to Psychoeducation for Smoking Precontemplators With SMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, A. Eden Evins, Director, Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: P2006
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Nicotine Dependence
Keywords: Transtheoretical Model; Stages of Change; Nicotine Dependence; Severe Mental Illness
MeSH Terms: conditions — Tobacco Use Disorder; Mental Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): The Cognitive Behavioral Therapy/Motivational Interviewing group consisted of four group sessions focused on using motivational interviewing to enhance motivation to quit smoking and on presenting cognitive-behavioral techniques for preparing to cut down or quit smoking. The following four topics were covered in this program: 1) Positive and Negative Aspects of Smoking, 2) Concerns and Hopes about Cutting Down or Quitting, 3) Small Changes that Can Help You Get Motivated, and 4) Planning for the Future.
  Interventions: Other: Motivational Interviewing
- Psychoeducation (Experimental): The education group also consisted of four group sessions that were co-led by a doctoral-level clinical psychologist and at bachelors-level research assistant. However, the focus of the education group was to present factual information about health risks of smoking, benefits of quitting, pharmacological smoking cessation aides, and smoking cessation programs in the area. The four group topics included: 1) Health Risks of Smoking, 2) Benefits of Quitting, 3) Nicotine Replacement Therapy and Bupropion (Zyban), and 4) Options for Treatment Programs.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Motivational Interviewing
  Arms: Motivational Interviewing
Other: Psychoeducation
  Arms: Psychoeducation

SUMMARY:
The investigators primary hypothesis was that recipients of the Motivational Interviewing intervention would be significantly more likely than those assigned to the Psychoeducation intervention to demonstrate increased readiness to quit smoking at the end of the intervention and to seek smoking cessation treatment in the one month period following the intervention. We also predicted that the Psychoeducation intervention would result in greater improvements in smoking knowledge.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Had a diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or chronic major depressive disorder by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria
* Smoked at least 10 cigarettes per day
* At baseline, reported not being ready to quit smoking within the next 30 days (i.e., in precontemplation or contemplation stages).

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Readiness to quit (Stage of Change) | 30 days
  efficacy of a cognitive behavioral therapy/motivational (MI) interviewing intervention relative to a psychoeducational (ED) intervention in terms of promoting increased readiness to quit smoking among smokers with severe mental illness who were not ready to quit.

SECONDARY OUTCOMES:
Smoking Knowledge | 30 days
  Changes in smoking knowledge obtained through cognitive behavioral therapy/motivational (MI) interviewing intervention relative to a psychoeducational (ED) intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Schizophrenia Program of the Massachusetts General Hospital, Freedom Trail Clinic, 25 Staniford St, Boston, Massachusetts, United States